CLINICAL TRIAL: NCT01833481
Title: In Vivo Determination of THA Kinematics and Sound for Subject Implanted Using Various Surgical Approaches
Brief Title: THA Kinematics and Sound for Subjects Implanted Using Various Surgical Approaches
Acronym: THA
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Other Study IDs: 12009; R01 1373 452 (Other: University of Tennessee); 13-0372 (Other: University of Tennessee)
Record Dates: First submitted 2013-04-11; First posted 2013-04-17 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Hip Injuries
Keywords: Surgical approach; Direct-anterior; Anterior-lateral; Posterior-lateral; Hip implant; Total Hip Arthroplasty; Total Hip replacement; Hip replacement; Hip prosthesis
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- THA using direct-anterior surgical approach: Patients will have undergone THA using a direct-anterior surgical approach and will undergo fluoroscopy surveillance while walking.
  Interventions: Radiation: Fluoroscopy surveillance of patients while walking
- THA using anterior-lateral approach: Patients will have undergone THA using an anterior-lateral surgical approach and will undergo fluoroscopy surveillance while walking.
  Interventions: Radiation: Fluoroscopy surveillance of patients while walking
- THA using posterior-lateral approach: Patients will have undergone THA using a posterior-lateral surgical approach and will undergo fluoroscopy surveillance while walking.
  Interventions: Radiation: Fluoroscopy surveillance of patients while walking

INTERVENTIONS:
Radiation: Fluoroscopy surveillance of patients while walking — While each subject performs a gait activity (normal walking) under fluoroscopic surveillance on a level treadmill, a data acquisition (DAQ) system will be used to determine the vibrations/sounds occurring during walking.
  Other Names: DePuy Orthopaedics hip implant

SUMMARY:
In a previous study conducted within the Center for Musculoskeletal Research (CMR) on Total Hip Arthroplasties (THA), it was determined that the investigators could simultaneously capture in vivo sound and motion of the femoral head within the acetabular cup during weight-bearing activities for subjects implanted with either a metal-on-polyethylene (MOP), metal-on-metal (MOM) or ceramic-on-ceramic (COC) THA. This was the first study to apply sound analysis as an impulse excitation technique for testing hip conditions and for measuring femoral head sliding in the acetabular component of human hip joints by acoustic means. Unfortunately, no studies have been conducted to compare the in vivo kinematics and sound for subjects implanted using various surgical approaches. It could be hypothesized that subjects having various surgical approaches could lead to an increase or reduction of in vivo hip separation. Therefore, the objective of this study is to analyze a total of 30 subjects implanted with either an anterior (10 patients), anterior-lateral (10 patients), or posterior-lateral (10 patients) surgical approach to determine if any of these surgical approaches leads to less or more in vivo hip separation. All subjects will be analyzed under in vivo weight-bearing conditions using video fluoroscopy to determine in vivo motion.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative clinical evaluation judged successful using Harris Hip Scoring (HHS) system (HHS>90)
* Body weight less than 270 lbs
* No evidence of post-operative hip subluxation or dislocation
* Do not walk with detectable limp
* Be able to actively abduct their operated hip against gravity without difficulty
* Must be willing to sign Informed Consent and Health Insurance Portability and Accountability (HIPAA) forms

Exclusion Criteria:

* Pregnant, lactating or females not using reliable form of birth control
* Patients that do not meet study requirements
* Patients unwilling to sign Informed Consent or HIPAA forms

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a direct-anterior surgical approach will be provided by Dr. William Barrett of Valley Orthopedic Associates in Renton, WA.
  Patients implanted with an anterior-lateral surgical approach will be provided by Dr. of Steven J. MacDonald of the London Health Sciences Center, London, Ontario.
  Patients implanted with a posterior-lateral approach will be provided by Dr. David F. Dalury of Towson Orthopaedic Associates, Inc. in Towson, MD.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Komistek, Ph D, Principal Investigator — The University of Tennessee; Adrija Sharma, Ph D, Principal Investigator — The University of Tennessee
Locations (3):
- United States (2):
  - University of Maryland St. Joseph Medical Center, Towson, Maryland
  - Valley Orthopedic Associates ASC, Renton, Washington
- University Hospital, London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | THA Using Direct-anterior Surgical Approach | THA Using Anterior-lateral Approach | THA Using Posterior-lateral Approach
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | THA Using Direct-anterior Surgical Approach | THA Using Anterior-lateral Approach | THA Using Posterior-lateral Approach | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (7.3) | 67 (5.4) | 69 (8.7) | 66 (7.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 3 | 12
  >=65 years | 4 | 7 | 7 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9 | 18
  Male | 5 | 6 | 1 | 12
Region of Enrollment [Number; unit: participants]
  United States | 10 | 0 | 10 | 20
  Canada | 0 | 10 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Kinematics - Swing Phase Separation
Description: Determine amount of in vivo swing phase hip separation present within implanted hip during weight-bearing level walking while under fluoroscopic surveillance.
Time Frame: 6 months post-operatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | THA Using Direct-anterior Surgical Approach | THA Using Anterior-lateral Approach | THA Using Posterior-lateral Approach
Number analyzed (Participants) | 10 | 10 | 10
mm | 0.9 (0.7) | 0.6 (0.3) | 1.0 (0.4)

2. Primary Outcome: Kinematics - Stance Phase Separation
Description: Determine amount of stance phase hip separation present in vivo of implanted hip during level walking activity under fluoroscopic surveillance.
Time Frame: 6 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | THA Using Direct-anterior Surgical Approach | THA Using Anterior-lateral Approach | THA Using Posterior-lateral Approach
Number analyzed (Participants) | 10 | 10 | 10
mm | 0.9 (0.3) | 0.8 (0.6) | 1.0 (0.3)

3. Primary Outcome: Kinematics - Overall Separation
Description: Determine overall hip separation present in vivo in implanted hip during level walking activity under fluoroscopic surveillance
Time Frame: 6 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | THA Using Direct-anterior Surgical Approach | THA Using Anterior-lateral Approach | THA Using Posterior-lateral Approach
Number analyzed (Participants) | 10 | 10 | 10
mm | 1.1 (0.6) | 0.8 (0.6) | 1.2 (0.4)

ADVERSE EVENTS:
Arm/Group | THA Using Direct-anterior Surgical Approach | THA Using Anterior-lateral Approach | THA Using Posterior-lateral Approach
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes